CLINICAL TRIAL: NCT06953193
Title: Intraoperative Hypotension in Pancreatoduodenectomy: A Randomized Trial of General Versus Combined Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Rafael Paulino Leal Villalpando, Chief of the Department of Anesthesiology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANE-4574-23-24-1
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Neoplasms; Hypotension; Pancreatoduodenectomy
Keywords: Pancreatic Surgery; General Anesthesia; Hemodynamic Changes; Vasopressors; Postoperative Complications; Combined Anesthesia
MeSH Terms: conditions — Pancreatic Neoplasms; Hypotension; Postoperative Complications | interventions — Anesthesia, General; Tea

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the investigator and the outcomes assessor will be blinded to the group assignment. Care providers will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Anesthesia (Active Comparator): Patients will receive general anesthesia for pancreatoduodenectomy. Standardized anesthetic technique will be used with induction and maintenance based on institutional protocols, including intravenous induction agents, inhalational anesthetics, and intraoperative monitoring. No epidural catheter will be placed.
  Interventions: Procedure: General Anesthesia
- Combined General Anesthesia (Thoracic Epidural) (Experimental): Patients will receive combined general anesthesia (thoracic epidural) for pancreatoduodenectomy. Standardized general anesthesia will be administered as in the general anesthesia group, with the addition of a thoracic epidural catheter placed before induction and maintained intraoperatively with local anesthetics according to institutional protocol.
  Interventions: Procedure: Combined General Anesthesia (Thoracic Epidural)

INTERVENTIONS:
Procedure: General Anesthesia — Patients will undergo balanced general anesthesia for pancreatoduodenectomy. Induction will include: fentanyl 4 mcg/kg, lidocaine 1 mg/kg, propofol 1.5 mg/kg, and rocuronium 0.6 mg/kg.
  Anesthesia maintenance will be achieved with sevoflurane (variable concentration as per anesthesiologist discretion) and continuous fentanyl infusion according to the attending anesthesiologist's judgment.
  No epidural catheter will be placed.
  Arms: General Anesthesia
Procedure: Combined General Anesthesia (Thoracic Epidural) — Patients will undergo combined general anesthesia (thoracic epidural) for pancreatoduodenectomy.
  Induction will include: fentanyl 4 mcg/kg, lidocaine 1 mg/kg, propofol 1.5 mg/kg, and rocuronium 0.6 mg/kg.
  A thoracic epidural catheter will be placed at the best palpable intervertebral space between T6-T9 by the attending anesthesiologist.
  Anesthesia maintenance will include sevoflurane (variable concentration), fentanyl infusion at the anesthesiologist's discretion, and continuous infusion of 0.25% bupivacaine via the epidural catheter throughout the surgery.
  Arms: Combined General Anesthesia (Thoracic Epidural)

SUMMARY:
This randomized clinical trial compares the hemodynamic effects of general anesthesia versus combined general anesthesia (thoracic epidural) in patients undergoing pancreatoduodenectomy. The primary aim is to assess the incidence of intraoperative hypotension and related adverse events. Secondary outcomes includes vasopressor requirements, transfusion needs, postoperative complications, intensive care unit admission, hospital length of stay, and mortality.

DETAILED DESCRIPTION:
Pancreatoduodenectomy is a major surgical procedure associated with significant hemodynamic challenges. Thoracic epidural anesthesia provides effective analgesia and may attenuate the surgical stress response, its intraoperative use has been associated with increased risk of hypotension and higher vasopressor requirements.

This randomized clinical trial aims to evaluate intraoperative hemodynamic changes in patients undergoing elective pancreatoduodenectomy managed with either general anesthesia or combined general anesthesia (thoracic epidural). A total of 206 patients will be enrolled at the "National Institute of Medical Sciences and Nutrition Salvador Zubirán". Patients will be randomized into two groups: one receiving general anesthesia and the other receiving combined general anesthesia (thoracic epidural).

Randomization will be performed using the REDCap platform with a simple 1:1 allocation ratio. Each patient's group assignment will be generated automatically by REDCap at the time of enrollment to ensure allocation concealment.

An independent observer, blinded to the anesthetic technique, will monitor and record episodes of hypotension throughout the perioperative period. The principal investigator will be blinded to group assignment.

Secondary outcomes include intraoperative vasopressor use, estimated blood loss, transfusion requirements, postoperative complications (such as pancreatic fistula, anastomotic leak, hemorrhage, surgical site infection, and acute kidney injury), admission to the intensive care unit, length of stay in the ICU and hospital, and mortality.

A planned interim analysis will be conducted after the enrollment of the first 66 patients to assess the safety and feasibility of the study protocol. Based on this analysis, modifications to improve patient safety may be recommended by the research team or ethics committee.

This study will help determine the optimal anesthetic strategy to minimize hemodynamic instability and postoperative morbidity in patients undergoing pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Patients scheduled for elective pancreatoduodenectomy at National Institute of Medical Sciences and Nutrition Salvador Zubirán.
* No contraindications for neuroaxial anesthesia (epidural catheter placement), including:

  * Generalized or localized infection at the puncture site.
  * Thrombocytopenia.
  * Coagulation disorders.
  * Intracranial hypertension.
  * Patient refusal.

Exclusion Criteria:

* Age under 18 years.
* Pregnancy.
* Inability to randomize the case due to specific circumstances (such as contraindications to epidural use), resulting in non-eligibility based on participation criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-01-07 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intraoperative Hypotension | From induction of anesthesia to end of surgery (intraoperative period).
  Defined as the occurrence of any mean arterial pressure (MAP) <65 mmHg during the intraoperative period, measured continuously with an invasive arterial line or intermittently with a non-invasive blood pressure monitor, as available.

SECONDARY OUTCOMES:
Type of Vasopressor Administered | From induction of anesthesia to end of surgery.
  Type of vasopressor administered intraoperatively, categorized as ephedrine, norepinephrine, adrenaline, dopamine, or dobutamine.
Estimated Blood Loss | From start to end of surgery.
  Total estimated intraoperative blood loss in milliliters.
Number of Blood Transfusions | From start to end of surgery.
  Number of units of packed red blood cells transfused intraoperatively.
ICU Admission Rate | Within 24 hours after surgery.
  Percentage of patients requiring admission to the intensive care unit after surgery.
Length of Hospital Stay | Up to 60 days after surgery
  Total number of days from the date of surgery to the date of hospital discharge.
Postoperative Complications | Up to 30 days after surgery.
  Incidence of postoperative complications such as pancreatic fistula, anastomotic leak, surgical site infection, hemorrhage, and acute kidney injury.
30-Day Mortality | 30 days postoperatively.
  All-cause mortality within 30 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No